CLINICAL TRIAL: NCT04928469
Title: Clinical Impact of Coronavirus Disease 19 (COVID-19) Caused by P.1 Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Lineage
Brief Title: Clinical Impact of COVID-19 by P.1 SARS-CoV-2 Lineage
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Principal Investigator, Alexandre Prehn Zavascki, Principal Investigator, Hospital de Clinicas de Porto Alegre
Other Study IDs: 2020-0163
Record Dates: First submitted 2021-06-13; First posted 2021-06-16 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Covid19; COVID-19 Pneumonia; SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — RT-PCR positive for SARS-CoV-2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- P.1: Patients infected with the P.1 SARS-CoV-2 variant
  Interventions: Other: No intervention performed
- Other variants: Patients infected with SARS-CoV-2 variants other than P.1
  Interventions: Other: No intervention performed

INTERVENTIONS:
Other: No intervention performed — Collection of clinical and laboratory data

SUMMARY:
Since the first report of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) variant of concern (VOC) P.1 in Manaus, Brazil, a rapid spread of this lineage across the country has been observed. Recent studies indicate that this variant is associated with higher transmissibility; it is not known whether it is associated with clinical severity and higher mortality rates.

This is a retrospective cohort study carried out at Hospital de Clínicas de Porto Alegre. Adult patients aged 18 years or more and 65 years or less who were admitted to the hospital due to symptomatic COVID-19 from June 2020 to May 2021 and had a reverse transcriptase-polymerase chain reaction (RT-PCR) cycle threshold value for either SARS-CoV-2 N1 or N2 target ≤ 25 were eligible to the study. Samples from 86 patients (43 from June 2020 to November 2020 and 43 from February 2021 to May 2021) were sequenced for further evaluation. These dates were defined since the emergence of P.1 lineage in late January.

Clinical data regarding ventilatory support, date of onset of symptoms, laboratory findings and mortality were collected from each patient. This retrospective cohort aims to assess whether the number of days needed for supplementary oxygen either by noninvasive ventilation or high-flow nasal cannula from onset of symptoms differs among patients infected with the P.1 SARS-CoV-2 variant and those infected with other variants.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years
* Hospital admission due to symptomatic COVID-19
* RT-PCR was collected from June to November 2020 or from February to May 2021

Exclusion Criteria:

* Patients admitted for reasons other than COVID-19
* Asymptomatic patients with positive routine screening with RT-PCR
* Patients transferred from other institutions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 65 years, seeking medical care in Hospital de Clínicas de Porto Alegre due to symptomatic COVID-19, admitted from June to November 2020 or from February to May 2021.
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Time to Advanced Respiratory Support | 28 days from onset of symptoms
  Number of days needed for supplementary oxygen either by noninvasive ventilation or high-flow nasal cannula from onset of symptoms.

SECONDARY OUTCOMES:
Proportion of patients in each category in the ordinal scale during hospitalization | 28 days from hospital admission
  Proportion of patients in each category in the ordinal scale during hospitalization. Ordinal scale levels: 1, patient not hospitalized; 2, hospitalized and not receiving supplemental oxygen; 3, hospitalized and receiving supplemental oxygen; 4, hospitalized and receiving oxygen supplementation administered by a high-flow nasal cannula or noninvasive ventilation; 5, hospitalized and receiving mechanical ventilation or extracorporeal membrane oxygenation; and 6, death.
Arterial oxygen partial pressure (PaO2)/ Fractional inspired oxygen (FiO2) evolution during hospitalization | 28 day from hospital admission
  Proportion of patients in each category according to PaO2/FiO2 value: 400-301, 300-201, 200-101, <=100.
28-day Mortality from onset of symptoms | 28 days from onset of symptoms
  Death for any cause from onset of symptoms
Time to death from onset of symptoms | 28 days from onset of symptoms
  Number of days from the onset of symptoms to death
28-day Mortality from hospital admission | 28 days from hospital admission
  Death for any cause from hospital admission
Time to death from hospital admission | 28 days from hospital admission
  Number of days from the hospital admission to death
Days alive and free of supplemental oxygen support. | 28 day from hospital admission
  Number of days alive and free of supplemental oxygen support
Time to invasive ventilatory support | 28 days from onset of symptoms
  Number of days from the onset of symptoms to mechanical ventilation or Extracorporeal membrane oxygenation (ECMO)
Need of critical care | 28 days from hospital admission
  Proportion of patients admitted to Intensive Care Unit
In-hospital mortality | 90 days from hospital admission
  Death for any cause during hospitalization
Number of thromboembolic event | 28 day from hospital admission
  Number of patients with documented deep venous thrombosis or pulmonary embolism
Number of patients requiring renal replacement therapy (RRT) | 28 day from hospital admission
  Number of patients requiring any form of RRT during hospitalization
Number of patients requiring prone positioning | 28 day from hospital admission
  Number of patients requiring prone positioning during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Statistical Analysis Plan — https://docs.google.com/document/d/11uN0slg6N6K_10vm4BuXVtB7_QcZOAf5M6P0I-okGkU/edit#